CLINICAL TRIAL: NCT03668275
Title: A Single-center, Open Randomized Controlled Clinical Trial to Evaluate the Quality and Cost of (Partial) Oncological Home-hospitalization Compared to Standard Ambulatory Hospital Care
Brief Title: Evaluating Quality and Cost of (Partial) Oncological Home-Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Koen Van Eygen, Head of Oncology, General Hospital Groeninge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AZGS2017075
Record Dates: First submitted 2017-08-16; First posted 2018-09-12 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): (partial) oncological home-hospitalization
  Interventions: Procedure: (partial) oncological home-hospitalization
- Control (No Intervention): standard oncological ambulatory hospital care

INTERVENTIONS:
Procedure: (partial) oncological home-hospitalization — Patients assigned to oncological home-hospitalization will receive as many as possible parts of their oncological treatment at their homes. These include the required preparatory actions before treatment administration is possible and/or the treatment administration itself in case of subcutaneous cancer drugs.
  Arms: Intervention

SUMMARY:
Oncological home-hospitalization might be a patient-centred, cost-effective approach to deal wiht the current challenges in cancer healthcare.

The primary aim of this clinical trial is to evaluate patient-reported quality of life of patients receiving (partial) oncological home-hospitalization and to compare this outcome with patients receiving standard ambulatory hospital care.

Secondary endpoints that will be evaluated and compared between both randomized groups are: Quality of life related endpoints (i.e. distress, depression & anxiety and general health-related quality of life); Costs; Safety; patients' reported Satisfaction & Preferences and Efficiency for the hospital day care unit.

ELIGIBILITY:
Inclusion Criteria:

* Starting new oncological treatment at the outpatient hospital
* ECOG ≤ 2
* Living within 30 minutes of drive from the hospital

Exclusion Criteria:

* Important comorbidity (ECOG > 2)
* Life expectancy < 6 months
* Simultaneous treatment with radiotherapy
* Taking part in clinical trial with any Investigational Medicinal Product
* Language barriers or communication difficulties
* Problematic venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient-reported Quality of Life - Cancer specific | Inquiry at baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluation of the change of patient-reported quality of life for both study arms using FACT-G (Functional Assessment of Cancer Therapy - General) questionnaire.
Change in Patient-reported Quality of Life - General | Inquiry at baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluation of the change of patient-reported quality of life for both study arms using EQ-5D (EuroQol 5 dimensions) questionnaire.

SECONDARY OUTCOMES:
Patient-reported Distress | Inquiry at baseline and 12 weeks
  Evaluation of distress for both study arms using Distress Barometer (DB).
Patient-reported Depression & Anxiety | Inquiry at baseline and 12 weeks
  Evaluation of depression and anxiety for both study arms using the hospital anxiety and depression scale (HADS).
Cost evaluation using study-specific costs questionnaire | 12 weeks
  Evaluation of healthcare use and related costs for both study arms, using a self-designed costs form in which patients can complete their healthcare use and related expenses during the course of the trial.
Number of grade 3/4 toxicities according to CTCAE v4.0 | Inquiry at baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluation of safety for both study arms, by registrating grade 3/4 toxicities (according to the CTCAE v4.0) during 12 weeks
Patient-reported Safety | Inquiry at baseline, 4 weeks, 8 weeks and 12 weeks
  Evaluation of patient-reported safety for both study arms, by assessing patients-reported feeling of safety using VAS (Visual analogue scale).
Satisfaction using OUT-PATSAT35 CT questionnaire | Inquiry at baseline and 12 weeks
  Evaluation of patients-reported satisfaction with the provided care in both study arms, using the Cancer Out-Patient Satisfaction with Care questionnaire (OUT-PATSAT35) .
Preference using a self-designed patient-reported questionnaire | Inquiry at baseline and 12 weeks
  Evaluation of patients-reported preference for the provided care in both study arms, using a self-designed preference questionnaire.
Wait times for administration of treatment at the oncology day care unit. | 12 weeks
  Evaluation of the efficiency of the workflow at the oncological day care unit for both study arms, by examining the waiting time for treatment administration for each visit of each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Az Groeninge, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No